CLINICAL TRIAL: NCT04857346
Title: Indocyanine-mediated Antimicrobial Photodynamic Therapy Promotes Superior Clinical Effects in Stage III and Grade C Chronic Periodontitis Among Different Forms of Diabetes Mellitus: A Randomized Controlled Clinical Trial
Brief Title: Antimicrobial Photodynamic Therapy in Chronic Periodontitis and Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mohammed Mahmoud Al-Momani, Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSU334
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus; Prediabetic State; Chronic Periodontitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Chronic Periodontitis | interventions — Indocyanine Green; Photochemotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controlled Type 2 diabetes mellitus (Experimental)
  Interventions: Drug: Indocyanine green
- Uncontrolled Type 2 diabetes melltius (Experimental)
  Interventions: Drug: Indocyanine green
- Non-diabetic patients (Active Comparator)
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Single application of PDT will be performed. A diode laser (HELBO®TheraLite - Bredent Medical, Germany) with 670 nm wavelength, power of 150 mW, fluency of 22 J/cm2 and density of 1.1 W/cm2 will be used in this study. Indocyanine-green photosensitizer (Sigm Aldrich, USA) with 0.005% concentration will be used as a photosensitizer which will be applied inside the periodontal pockets in a depth of 3 mm with the help of a blunt needle for 10 s. Laser irradiation will be performed for 60 s using a flexible tip. Laser irradiation will be performed at 2 points each on buccal and lingual with the tip stabilized perpendicular to the gingival tissues.
  Other Names: Photodynamic therapy

SUMMARY:
With this design, this study hypothesizes that; (i) ICG-PDT would produce superior clinical, microbiological, and immune-inflammatory outcomes as compared to RSD and (ii) ICG-PDT would produce equal efficacy among different forms of diabetes as produced in non-diabetic subjects and that diabetes mellitus would not produce negative impact on the therapeutic outcomes of ICG-PDT. Therefore, the aim of this randomized controlled clinical trial was to evaluate the efficacy of ICG-mediated aPDT in the treatment of stage III grade C periodontitis among patients with prediabetes, T2DM and non-diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥30 years
2. clinically diagnosed with mild to moderate periodontitis
3. self-reported type-2 DM for ≥2 years confirmed by a physician with HbA1c levels ≥6.5%
4. patients who complied with the treatment protocol.

Exclusion Criteria:

(i) pregnancy and lactation (ii) who had taken antibiotics in the previous 3 months (iii) who had undergone periodontal therapy or any decontamination treatment in their oral cavity in the previous 6 months (iv) former/current smokers (v) failure to provide a signed informed consent.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Probing depth | 6 months
  Probing depth will be measured to the nearest millimeter from the base of the periodontal pocket to the crest of the marginal gingiva.
Clinical attachment level | 6 months
  Clinical attachment level will be measured by adding recession with probing depth

SECONDARY OUTCOMES:
Plaque scores | 6 months
  Dichotomous scoring to each site of the tooth as '1 - present' and '0 - absent'
Bleeding on probing | 6 months
  Dichotomous scoring to each site of the tooth as '1 - present' and '0 - absent'
Porphyromonas gingivalis | 6 months
  Presence or absence of bacteria from the plaque biofilms in the patient
Interleukin-6 | 6 months
  Proinflammatory cytokine levels that will be quantified in the laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Applied Medical Sciences, King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Momani MM. Indocyanine-mediated antimicrobial photodynamic therapy promotes superior clinical effects in stage III and grade C chronic periodontitis among controlled and uncontrolled diabetes mellitus: A randomized controlled clinical trial. Photodiagnosis Photodyn Ther. 2021 Sep;35:102379. doi: 10.1016/j.pdpdt.2021.102379. Epub 2021 Jun 1. PMID 34087466